CLINICAL TRIAL: NCT01149850
Title: Phase II Study of Bevacizumab and Temozolomide in Elderly Patients With Newly-Diagnosed Glioblastoma
Brief Title: Bevacizumab and Temozolomide in Treating Older Patients With Newly-Diagnosed Glioblastoma Multiforme or Gliosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-000760; AVF4535s (Other: UCLA IRB); 09-06-032 (Other: UCLA IRB)
Record Dates: First submitted 2010-06-22; First posted 2010-06-24 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Giant Cell Glioblastoma; Glioblastoma; Gliosarcoma
Keywords: adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Bevacizumab; Temozolomide; Immunohistochemistry; Microarray Analysis; Gene Expression Profiling; DNA Methylation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm I (Experimental): Patients receive bevacizumab IV over 30-90 minutes every 2 weeks and oral temozolomide on days 1-5. Treatment repeats every 28 days for 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: temozolomide; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: microarray analysis; Genetic: DNA methylation analysis

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; anti-VEGF rhuMAb; Avastin; recombinant humanized anti-VEGF monoclonal antibody; rhuMAb VEGF
Drug: temozolomide — Given orally
  Other Names: CCRG-81045; M & B 39831; SCH 52365; Temodal; Temodar; TMZ
Other: laboratory biomarker analysis — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: microarray analysis — Correlative studies
  Other Names: gene expression profiling
Genetic: DNA methylation analysis — Correlative studies

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as temozolomide, also work in different ways to kill tumor cells or stop them from growing. Giving bevacizumab together with temozolomide may be a better way to block tumor growth.

PURPOSE: This phase II trial is studying how well giving bevacizumab and temozolomide together works in treating older patients with newly diagnosed glioblastoma multiforme or gliosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate overall survival in elderly subjects treated with bevacizumab and temozolomide for newly diagnosed glioblastoma multiforme.

SECONDARY OBJECTIVES:

I. To estimate 12-months survival. II. To estimate progression free survival for 2 years or until progression is detected.

III. To investigate the safety and tolerability of bevacizumab/temozolomide in elderly patient with glioblastoma.

IV. To isolate DNA, RNA, and protein isolated from frozen and paraffinized archival tumor samples for evaluations such as immunohistochemical pathway profiling of VEGF-dependent angiogenic pathways, gene expression microarray, and MGMT promoter methylation status to define important molecule features of treatment response and especially age-related molecular expression.

OUTLINE:

Patients receive bevacizumab IV over 30-90 minutes every 2 weeks and oral temozolomide on days 1-5. Treatment repeats every 28 days for 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at least every 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have histologically proven intracranial glioblastoma multiforme (GBM) or gliosarcoma (GS); this includes treatment-naive patients with prior tissue diagnosis of lower grade gliomas that have been upgraded after repeat resection
* Cranial MRI or contrast CT must have been performed within 21 days of study entry; the use of MRI rather than CT is preferred; the same type of scan, i.e., MRI or CT, must be used throughout the period of protocol treatment for tumor measurement; if the surgical procedure was a resection, cranial MRI or contrast CT performed within 96 hours of resection is preferred, but not required; patients without measureable or assessable disease are eligible
* Patients must begin temozolomide chemotherapy no sooner than 2 weeks and no later than 6 weeks from the diagnostic surgery; patients must begin bevacizumab no sooner than 4 weeks and no later than 6 weeks from the surgery
* Patients must be willing to forego other drug therapy against the tumor while being treated with bevacizumab and temozolomide
* All patients must sign and informed consent approved by the Institutional Review Board indicating that they are aware of the investigational nature of this study; patients must also sign an authorization for the release of their protected heath information
* Life expectancy > 8 weeks
* Patients must have a Karnofsky performance status of >= 60
* WBC >= 3,000/ul
* ANC >= 1,500/mm^3
* Platelet count of >= 100,000/mm^3
* Hemoglobin >= 10 gm/dl
* SGOT < 2.5 times ULN
* Bilirubin < 2.5 ULN
* Patients must have adequate renal function (creatinine < 1.5 mg/dL) before starting therapy and the test must be performed within 14 days prior to registration

Exclusion Criteria:

* Glioblastoma disease-specific concerns: Patients must not have received previous or concurrent radiotherapy to the brain
* Glioblastoma disease-specific concerns: Patients must have received cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy directed against the brain tumor; patients who received Gliadel wafers will be excluded; patients may have received or be receiving corticosteroids, AED's, analgesics, and other drugs to treat symptoms or prevent complications
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Patients with a history of any other cancer (except non-melanoma skin cancer, carcinoma in-situ of the cervix, or low-risk prostate cancer after curative therapy), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible
* Patients receiving current, ongoing treatment with full-dose warfarin or its equivalent (i.e., unfractionated and/or low molecular weight heparin) are NOT excluded
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism
* Patients must not have serious uncontrolled inter-current medical illness including, but not limited to, ongoing or active infection requiring IV antibiotics, psychiatric illness/social situations that would limit compliance with study requirements, or disorders associated with significant immunocompromised state (HIV, SLE, etc.)
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Blood pressure of > 150/100 mmHg, history of hypertensive crisis or hypertensive encephalopathy
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months prior to day 1
* History of stroke within 6 months prior to day 1
* International normalized ratio (INR) > 1.5 and activated partial thromboplastin time (aPTT) > 1.5 x the ULN (except for subjects receiving anticoagulation therapy) in the absence of therapeutic intent to anticoagulate the subject; therapeutic anticoagulation is permitted
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis ( >= 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury other than craniotomy within 28 days prior to Day 1, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as placement of Port-a-Cath, stereotactic biopsy, fine needle aspirations, or core biopsies within 7 days prior to Day 1
* History of intracerebral abscess within 6 months prior to Day 1
* Urine protein: creatinine ratio >= 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1
* Serious, non-healing wound, ulcer, or bone fracture; patients with any wound requiring surgical intervention (including scalp wounds requiring cranioplasty) will be allowed to resume the study if the wound is clean and without further infection post-surgical intervention
* Known hypersensitivity to any component of bevacizumab
* Inability to comply with study and/or follow-up procedures

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-04-28 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Pts who progress followed for survival every 4 mths.Pts completing therapy & no progression followed every 2 mths/12 mths,every 3 mths/12 mths,every 4 mths/12 mths,every 6 mths until progression,then followed every 4 mths for survival

SECONDARY OUTCOMES:
Time to progression | 2 years
  Pts who progress followed for survival every 4 mths.Pts completing therapy & no progression followed every 2 mths/12 mths,every 3 mths/12 mths,every 4 mths/12 mths,every 6 mths until progression.
progression free survival | 2 years
  Patients completing therapy & no progression followed every 2 mths/12 mths,every 3 mths/12 mths,every 4 mths/12 mths,every 6 mths until progression,then followed every 4 mths for survival

CONTACTS AND LOCATIONS:
Overall Officials: Phioanh Nghiemphu, Principal Investigator — University of California at Los Angeles (UCLA )
Locations (3):
- United States (3):
  - Kaiser Foundation Hospital, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Kaiser Permanente at San Diego, San Diego, California